CLINICAL TRIAL: NCT02913846
Title: The Impact of Denutrition on the Hospital Length of Stay for Patients Undergoing Rehabilitation
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Samar Hatem, Head of clinic, Brugmann University Hospital
Other Study IDs: CHUB-Nut-Reva
Record Dates: First submitted 2016-09-14; First posted 2016-09-26 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Denutrition
Keywords: denutrition; hospital length of stay; patient's autonomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospital revalidation units: The study will take place within the CHU Brugmann hospital (Brussels) who has 4 revalidation units (104 beds). All patients coming within these units during the study duration will be included.
  Interventions: Other: Nutritional evaluation; Other: Muscular assessment; Other: Pre-albumine dosage

INTERVENTIONS:
Other: Nutritional evaluation — A first nutritional evaluation will be performed within 48h of patient admission. Weight and BMI will be measured once a week.
Other: Muscular assessment — An assessment of muscular force will be performed once a week.
Other: Pre-albumine dosage — Dosage performed once a month.

SUMMARY:
Denutrition is defined as a measurable decrease in functions and/or as change in the body composition, associated with a worsening of the prognosis of the underlying medico-surgical pathology. It is induced by a deficiency in energy, proteins or any other micro or macronutrient and is the result of malnutrition, itself caused by a poor diet or a metabolic disorder.

According to the National Nutrition and Health Plan for Belgium, denutrition is an independent risk factor for the increase of complications, morbidity and mortality rates, average length of hospitalisation and global medical care cost. It is necessary to invest in the prevention of denutrition as the costs of preventive measures are lower than the cost of treating a denutrished patient.

The Belgian financing system of hospitalisation days is based on the structure of the treated pathologies, the age of the patient and the geriatric features of the patient. It encourages all hospitals to lower the length of hospitalisation to the national average for all these criteria. As a consequence, there is a mounting tendency to shorten the average length of stay within the hospital.

The so-called 'Sp' hospital departments occupy a specific place within the organisation of Health Services in Belgium. They are specialized in the treatment and rehabilitation of patients with cardiopulmonary, neurological, locomotor, psycho-geriatric and chronic diseases. These services act as an extension of acute services (continuity of acute hospitalisation) but also as a first entry point for the medical care of patients with various specific diseases (multiple sclerosis, psycho-geriatric disorders, chronic pulmonary disorders...).

The financing of the Sp departments is, as opposed to the financing of other departments, not linked to the patient length of stay. However, an increase in hospitalization duration decreases the rate of admissions and the possibility to accept patients coming from acute hospital units.

The aim of the study is to evaluate the influence of denutrition of patients hospitalized in an Sp department on the length of revalidation stay, the associated costs and the patient's functional autonomy.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted within a revalidation unit of the CHU Brugmann hospital

Exclusion Criteria:

* Patients without programmed exit: transfer to another care unit, forced exit, death...

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted within a revalidation unit of the CHU Brugmann hospital
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2016-03-18 (Actual); Primary Completion 2017-09-12 (Actual); Study Completion 2017-09-12 (Actual)

PRIMARY OUTCOMES:
Barthel index score | within 48h of admission within the revalidation unit
  Assessment of patient autonomy
Nutritional Risk Screening score | within 48h of admission within the revalidation unit
  Nutritional state assessment
Body Mass Index | once a week up to patient discharge (the average hospitalization length within the revalidation unit is 48 days)
Weight | once a week up to patient discharge (the average hospitalization length within the revalidation unit is 48 days)
Hand prehension force | once a week up to patient discharge (the average hospitalization length within the revalidation unit is 48 days)
  performed on the right hand with a Jamart dynamometer
Pre-albumine level (mg/l) | once a week up to patient discharge (the average hospitalization length within the revalidation unit is 48 days)
  Laboratory testing

CONTACTS AND LOCATIONS:
Overall Officials: Samar Hatem, MD, Study Director — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alvarez-Hernandez J, Planas Vila M, Leon-Sanz M, Garcia de Lorenzo A, Celaya-Perez S, Garcia-Lorda P, Araujo K, Sarto Guerri B; PREDyCES researchers. Prevalence and costs of malnutrition in hospitalized patients; the PREDyCES Study. Nutr Hosp. 2012 Jul-Aug;27(4):1049-59. doi: 10.3305/nh.2012.27.4.5986. PMID 23165541